CLINICAL TRIAL: NCT02799368
Title: A Randomized, Open Label, Active Control, 2 Parallel Groups, Multicenter, Phase III Study to Evaluate the Efficacy and Safety of Balanced Salt Solution Versus 0.9% Saline in Patients With High Risk of Contrast Induced Nephropathy.
Brief Title: Balanced Salt Solution Versus 0.9% Saline Infusion for Prevention of Contrast-induced Acute Kidney Injury (BASIC Trial)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Kyungpook National University Hospital (Other); National Medical Center, Seoul (Other); National Health Insurance Service Ilsan Hospital (Other); Seoul National University Bundang Hospital (Other); Bundang CHA Hospital (Other); Seoul St. Mary's Hospital (Other); Seoul National University Boramae Hospital (Other); Severance Hospital (Other); Ewha Womans University Mokdong Hospital (Other); Incheon St.Mary's Hospital (Other); Gachon University Gil Medical Center (Other)
Responsible Party: Principal Investigator, Kwon wook Joo, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BS-CCT-01
Record Dates: First submitted 2016-06-10; First posted 2016-06-14 (Estimated); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Acute Kidney Injury; Renal Insufficiency, Chronic; Contrast Media Reaction
MeSH Terms: conditions — Acute Kidney Injury; Renal Insufficiency, Chronic | interventions — Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CJ Plasma Solution A Injection (Experimental): Before contrast media administration : CJ Plasma Solution A Injection (3mL/kg for 1 hour) After contrast media administration : CJ Plasma Solution A Injection (1.5 mL/kg/h for 4 hours)
  Interventions: Drug: CJ Plasma Solution A Injection
- CJ 0.9% Normal Saline Injection (Active Comparator): Before contrast media administration : CJ 0.9% Normal Saline Injection (3mL/kg for 1 hour) After contrast media administration : CJ 0.9% Normal Saline Injection (1.5mL/kg/h for 4 hours)
  Interventions: Drug: CJ 0.9% Normal Saline Injection

INTERVENTIONS:
Drug: CJ Plasma Solution A Injection — Intravenous plasma solution (Chloride 90 mmoL/L) at 3 mL/kg over 1 hour pre-contrast, followed by the same solution intravenously at 1.5 mL/kg/hr for 4 hours. Intra-vascular low-osmolal or iso-osmolal contrast will be used.
  Arms: CJ Plasma Solution A Injection
Drug: CJ 0.9% Normal Saline Injection — Intravenous plasma solution (Chloride 154 mmoL/L) at 3 mL/kg over 1 hour pre-contrast, followed by the same solution intravenously at 1.5 mL/kg/hr for 4 hours. Intra-vascular low-osmolal or iso-osmolal contrast will be used.
  Arms: CJ 0.9% Normal Saline Injection

SUMMARY:
As iodinate contrast media (CM) has been widely used in current medical practice, contrast induced acute kidney injury (CI-AKI) has been an important issue.

Previously, many guidelines suggested prophylaxis protocol using 0.9% saline when CM is administrated to high risk patients. However, recent studies showed that 0.9% saline might induce metabolic acidosis due to its supra-physiologic chloride component, and therefore renal vasoconstriction. In spite of protective effect by volume expansion with saline infusion, this renal vasoconstriction might have conflicting effect on renal function, as hypoxic injury is suspected to be the main cause of CI-AKI.

In contrast to 0.9% saline, balanced salt solution has physiologic level of chloride and neutral pH. Also, recent studies proved preventive effect of balanced salt solution for AKI in several clinical settings.

Hence, the investigators planned a prospective randomized controlled trial comparing 0.9% saline and balanced salt solution to prevent CI-AKI.

DETAILED DESCRIPTION:
Iodinated contrast media (CM) has been widely used for various diagnostic and therapeutic interventions. Coronary angiography and contrast enhanced computed tomography are representative medical procedure in which CM administration is necessary, and their usage are recently extended. Also, U.S sales of medical imaging CM has been increased.

Although iodinated CM has useful role in many medical procedures, CM is well known for its renal side effect, contrast induced acute kidney injury (CI-AKI). CI-AKI is one of the leading cause of iatrogenic acute kidney injury (AKI). Moreover, CI-AKI is known to be an independent risk factor for short- and long term morbidity and mortality. Considering the current rising incidence of CI-AKI, its prevention has been an important issue.

The incidence of CI-AKI is below 5% and up to 25% according to presence of risk factors such as renal failure, diabetes mellitus, heart failure, old age and concomitant use of nephrotoxic medications. Chronic kidney disease (CKD) is an established risk factor for CI-AKI and therefore several guidelines recommend prophylaxis for CI-AKI when patients with creatinine clearance (CrCl) below 60mL/min receives CM administration. In those guidelines, it is generally recommend that high risk patients should receive isotonic crystalloid solution and be considered for taking N-acetylcysteine, although there are still debates on its benefit.

Several clinical studies have compared 0.9% saline and sodium bicarbonate solution for their effectiveness on CI-AKI prevention, and no superiority was shown in using sodium bicarbonate solution. Hence, most organization currently use 0.9% saline for CI-AKI prophylaxis due to its wide availability.

However, several studies showed that 0.9% saline has supra-physiologic dose of chloride and induces metabolic acidosis which contributes renal vasoconstriction and impairment of estimated glomerular filtration rate (eGFR). Double blind, randomized clinical human study proved that these problems are less pronounced with the use of balanced salt solution, which has physiologic level of chloride and neutral pH. Also, recent prospective pilot study suggested that using chloride restrictive solutions, rather than using chloride rich solutions, for fluid resuscitation in critically ill patients can reduce AKI. Considering the above findings, few large scale cohort studies and randomized controlled trials are ongoing to prove preventive effect of balanced salt solution for AKI over 0.9% saline.

In conclusion, as stated above, use of 0.9% saline for CI-AKI prophylaxis might have limited benefit only by volume expansion. Considering its components, additional physiologic advantage by using balanced salt solution could be achieved. In order to assess this hypothesis, the investigators planned a multicenter prospective randomized controlled open-label trial comparing balanced salt solution and 0.9% saline to prevent CI-AKI.

The primary end-point of this study is event of CI-AKI, which is defined by relative (≥25%) or fixed (≥0.5mg/dL) increase in serum creatinine from baseline value assessed at 48 hours after CM use. The secondary end-point are decrease in eGFR of more than 50% from the baseline eGFR within 48 hours and initiation of dialysis and mortality, after 1 or 6 month from CM exposure. For this purpose, at least 830 subjects would be required for each group when type I error rate is 2.5% and type II error is 20%, given 20% drop-out rate during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18 years or older
* with eGFR < 45 mL/min/1.73m2 or eGFR < 60 mL/min/1.73m2 who have at least one condition Diabetes mellitus Age > 60 year
* Able and willing to provide informed consent

Exclusion Criteria:

* eGFR < 15 mL/min/1.73m2 or end stage renal disease patients with dialysis history
* Heart failure with left ventricular ejection fraction < 45% or severe symptoms (New York Heart Association functional classification III or IV)
* Decompensated heart failure patients who use dobutamine, dopamine, milrinone, amrinone, nesiritide or patients who have acute pulmonary edema
* History of hyperkalemia (serum K > 5.5 mEq/L) or hypernatremia ( serum Na > 145 mEq/L) in screening period
* Recent exposure to radiocontrast within 7 days of the study
* History of hypersensitivity to radiocontrast
* Multiple myeloma
* Pregnant/lactation
* Expected survival < 6 months
* Enrolled in other clinical trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 493 (Actual)
Dates: Start 2016-11; Primary Completion 2019-05 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Contrast Induced Acute Kidney Injury | 0-48 hour
  Relative (≥25%) or fixed (≥0.5mg/dL) increase in serum creatinine

SECONDARY OUTCOMES:
Decrease in renal function | 0-48 hour
  Decrease in eGFR of more than 50% from the baseline eGFR
1 month Renal replacement therapy | 0 to 30 days
  Initiation of renal replacement therapy
6 month Renal replacement therapy | 0 to 180 days
  Initiation of renal replacement therapy
1 month Mortality | 0 to 30 days
  Mortality
6 month Mortality | 0 to 180 days
  Mortality
Acute Kidney Injury by KDIGO guideline after CT scan | 0-48 hour
  Relative (≥50%) or fixed (≥0.3mg/dL) increase in serum creatinine (otherwise specified in the latest release of KDIGO guideline)

CONTACTS AND LOCATIONS:
Overall Officials: Kwon-Wook Joo, MD, PhD, Study Chair — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Park S, Kim DK, Jung HY, Kim CD, Cho JH, Cha RH, Jeong JC, Kim S, Kim HJ, Ban TH, Chung BH, Lee JP, Park JT, Han SH, Yoo TH, Ryu DR, Moon SJ, Lee JE, Huh W, Kang EW, Chang TI, Joo KW. Efficacy and Safety of a Balanced Salt Solution Versus a 0.9% Saline Infusion for the Prevention of Contrast-Induced Acute Kidney Injury After Contrast-Enhanced Computed Tomography. Kidney Med. 2020 Feb 21;2(2):189-195. doi: 10.1016/j.xkme.2019.12.003. eCollection 2020 Mar-Apr. PMID 32734238
- [Derived] Jo HA, Park S, Kim CD, Jung HY, Cho JH, Cha RH, Kang EW, Chang TI, Kim S, Kim HJ, Chung BH, Lee JP, Park JT, Han SH, Yoo TH, Ryu DR, Moon SJ, Chang JH, Kim DK, Joo KW. Efficacy and safety of a balanced salt solution versus a 0.9% saline infusion for the prevention of contrast-induced acute kidney injury (BASIC trial): a study protocol for a randomized controlled trial. Trials. 2017 Oct 5;18(1):461. doi: 10.1186/s13063-017-2202-2. PMID 28982378